CLINICAL TRIAL: NCT06625931
Title: A Randomized, Open-labeled, Multi-center, Active-controlled, Parallel-group Phase 3 Clinical Trial to Evaluate the Safety and Efficacy of NTCB01-1 Versus NTCB-P in Patients Who Require Parenteral Nutrition
Brief Title: Clinical Trial to Evaluate the Safety and Efficacy of NTCB01-1 in Patients Who Require Parenteral Nutrition
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NTCB01-301
Record Dates: First submitted 2024-10-02; First posted 2024-10-03 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-01

CONDITIONS: Parenteral Nutrition
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NTCB01-1 (Experimental)
  Interventions: Drug: NTCB01-1
- NTCB-P (Active Comparator)
  Interventions: Drug: NTCB-P

INTERVENTIONS:
Drug: NTCB01-1 — 3 Days infusion
  Arms: NTCB01-1
Drug: NTCB-P — 3 Days infusion
  Arms: NTCB-P

SUMMARY:
A Randomized, Open-labeled, Multi-center, Active-controlled, Parallel-group Phase 3 Clinical Trial to Evaluate the Safety and Efficacy of NTCB01-1 versus NTCB-P in patients who require parenteral nutrition

ELIGIBILITY:
Inclusion Criteria:

* Those who are 19 years old or older at the screening visit
* Patients are expected to require PN for more than 3 days
* Patients who voluntarily signed the consent form

Exclusion Criteria:

* Patients are expected difficult to survive more than 3 days
* Patients BMI is over 30 kg/m2
* Patients having hypersensitivity to any peanut-, fish-, soy-, egg protein, or investigational drug
* Patients with difficult peripheral intravenous line
* Patients judged to be unsuitable for this trial by investigators

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Occurance rate of adverse drug reaction | Day 1 to day 4

CONTACTS AND LOCATIONS:
Locations (7):
- South Korea (7):
  - Keimyung University Dongsan Hospital, Daegu, Dalseo-gu
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, Dongjak-gu
  - Seoul National University Hospital, Seoul, Jongno-gu
  - Kosin University Gospel Hospital, Busan, Seo-gu
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul, Seocho-Gu
  - Korea University Anam Hospital, Seoul, Seongbuk-gu
  - Ajou University Medical Center, Gyeonggi-do, Suwon-si

IPD SHARING:
Plan to Share IPD: No